CLINICAL TRIAL: NCT04575363
Title: RPSA as a Potential Prognostic Biomarker of PDAC
Brief Title: RPSA as a Potential Prognostic Biomarker of Pancreatic Cancer
Acronym: PaCaBioMarkeR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA20113
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
Keywords: Pancreatic ductal adenocarcinoma; Ribosomal protein SA (RPSA); prognosis biomarker
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pancreatic adenocarcinoma patient (Experimental): patient with pancreatic ductal adenocarcinoma
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample

SUMMARY:
PDAC (Pancreatic ductal adenocarcinoma) represents 90% of pancreatic tumors. The prognosis of PDAC remains poor at this time. Its management is based on surgery for early stages, associated with neoadjuvant and adjuvant chemotherapy. However, around 80% of patients will relapse after surgery. There is a lack of efficient biological biomarkers of PDAC, especially for prognosis. To date, CA19-9 is commonly used despite its lack of sensitivity and specificity.

Ribosomal protein SA (RPSA) is a transmembrane receptor localized at the cell surface but also in the cytosolic and nuclear regions. RPSA interacts with many proteins in the extracellular matrix (ECM), including laminin-1 and elastin. RPSA in involved in different cellular functions such as cell adhesion, migration, proliferation and differentiation. The expression of RPSA is increased in many cancers including breast, lung, prostate, pancreatic, etc. It could represent a molecular biomarker of tumor invasion and metastatic abilities. Moreover, the concentration of RPSA could be measured in the serum of patients with PDAC. Recent data suggest that a modification of the RPSA concentration could be a prognostic biomarker of PDAC.

DETAILED DESCRIPTION:
The aim of this study is to explore the potential implication of RPSA as prognostic biomarker of PDAC.

ELIGIBILITY:
inclusion criteria :

* Patients treated at the Reims University Hospital for a resectable or potentially resectable pancreatic tumor, with or without neoadjuvant chemotherapy
* Adults (aged more than 18 years old)
* Patients who have signed the informed consent form

exclusion criteria :

* Patients with a prior history of cancer (excluding basal cell carcinoma or in situ cervical cancer that received conventional cancer treatment).
* Minors
* Patients for whom PDAC is not the retained diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2026-10-18 (Estimated); Study Completion 2027-10-18 (Estimated)

PRIMARY OUTCOMES:
RPSA serum concentration | Day 0
  The RPSA serum concentration is assessed with commercially available RPSA ELISA assay (MyBioSource - MBS9137288).

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France